CLINICAL TRIAL: NCT01564563
Title: A Multi-center, Randomized, Double-blind, Parallel Groups, Placebo-controlled Trial on Efficacy and Safety of Activated Recombinant Factor VII (rFVIIa/NovoSeven®) in the Treatment of Bleeding in Patients Following Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Efficacy and Safety of Activated Recombinant Human Factor VII in Treatment of Bleeding in Patients Following Hematopoietic Stem Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial enrollment was prematurely terminated due to excessively slow patient recruitment
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7SCT-1485
Record Dates: First submitted 2012-03-23; First posted 2012-03-28 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Acquired Bleeding Disorder; Bleeding During/Following Surgery
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: standard therapy; Drug: placebo
- Low dose (Experimental)
  Interventions: Drug: standard therapy; Drug: activated recombinant human factor VII
- High dose (Experimental)
  Interventions: Drug: standard therapy; Drug: activated recombinant human factor VII

INTERVENTIONS:
Drug: standard therapy — Standard treatment of bleeding
Drug: placebo — Placebo
  Arms: Placebo
Drug: activated recombinant human factor VII — Two days repeated treatment regimen - low dose administered i.v. (into the vein)
  Arms: Low dose
Drug: activated recombinant human factor VII — Two days repeated treatment regimen - high dose administered i.v. (into the vein)
  Arms: High dose

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to evaluate the efficacy of activated recombinant human factor VII in treatment of bleeding in patients having undergone a hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone a hematopoietic stem cell transplantation

Exclusion Criteria:

* Known or suspected allergy to trial product
* Participation in other trials with unapproved drugs or trials with equal or similar objective

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2002-06-28 (Actual); Primary Completion 2003-10-27 (Actual); Study Completion 2003-10-27 (Actual)

PRIMARY OUTCOMES:
Effect on bleeding, defined as change in bleeding score

SECONDARY OUTCOMES:
Transfusion requirements
Bleeding evaluation
Adverse events
Changes in safety coagulation parameters

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (7):
- United States (7):
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, Duarte, California
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Houston, Texas

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com